CLINICAL TRIAL: NCT02611752
Title: A Multiple Dose Opioid Challenge Study to Assess Blockade of Subjective Opioid Effects of CAM2038 q1w (Buprenorphine FluidCrystal® Subcutaneous Injection Depots) In Adults With Opioid Use Disorder
Brief Title: A Multiple Dose Opioid Challenge Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-13-478
Record Dates: First submitted 2015-11-18; First posted 2015-11-23 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2018-08

CONDITIONS: Moderate or Severe Opioid Use Disorder
MeSH Terms: conditions — Lymphoma, Follicular; Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAM2038 q1w, 24 mg (Experimental): CAM2038 q1w 24 mg will be administered on Day 0 and Day 7. Hydromorphone 0 mg (placebo), 6 mg and 18 mg will be subsequently administered during 4 challenge sessions on Days 1-3, 4-6, 8-10 and 11-13
  Interventions: Drug: CAM2038
- CAM2038 q1w, 32 mg (Experimental): CAM2038 q1w 32 mg will be administered on Day 0 and Day 7. Hydromorphone 0 mg (placebo), 6 mg and 18 mg will be subsequently administered during 4 challenge sessions on Days 1-3, 4-6, 8-10 and 11-13
  Interventions: Drug: CAM2038

INTERVENTIONS:
Drug: CAM2038 — CAM2038 subcutaneous injection

SUMMARY:
Multi-site, randomized, double-blind, repeat-dose Phase 2 study to evaluate the degree and duration of action of multiple doses of CAM2038 in blocking the effects of hydromorphone in patients with moderate or severe opioid use disorder.

DETAILED DESCRIPTION:
This is a multi-site, randomized, double-blind, repeat-dose Phase 2 study to evaluate the degree and duration of action of multiple doses of CAM2038 q1w in blocking the effects of a mu opioid agonist (hydromorphone) in patients with moderate or severe opioid use disorder. The study will involve 4 phases: Screening, Qualification, Treatment, and Follow-up.

The study will enroll a sufficient number of subjects to ensure that at least 48 subjects complete the study (24 subjects per group with at least 16 females in total). Replacement subjects may be added at the discretion of the sponsor with the agreement of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patient had to provide written informed consent prior to the conduct of any study-related procedures.
2. Male or female, 18-55 years of age, inclusive.
3. Patients with a diagnosis of moderate or severe opioid use disorder (DSM-V) who were physically dependent on intravenous (IV) or insufflated opioids, and who were willing to undergo short-term BPN treatment.
4. Self-reported opioid-use of a minimum of 21 days in the 30 days prior to Screening.
5. Positive UDS for opioids at Screening or at check-in. If UDS was not positive, patients had to present with physical signs of withdrawal, as determined by the Investigator. The Investigator may have administered a naloxone challenge, in order to confirm opioid dependence at the Investigator's discretion.
6. Female patients of childbearing potential had to be willing to use a reliable method of contraception during the entire study (Screening Visit to Follow-up Phone Call).
7. Female patients of non-childbearing potential were surgically sterile (i.e., had undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels.
8. Male patients with female partners of childbearing potential had to agree to use a reliable method of contraception from Screening Visit through at least 3 months after the last dose of study drug. Male patients also must have agreed not to donate sperm during the study through at least 3 months after the last dose of study drug.
9. Were willing and able to comply with the study requirements (including blood sampling), complete study assessments, visit the clinic, and remain confined in the CRU for up to 25 consecutive days.

Exclusion Criteria:

1. History or presence of any clinically significant psychiatric, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or other major disease or illness at Screening, which in the opinion of the Investigator would have jeopardized the safety of the patient or the validity of the study results.
2. Opioid-dependent patients who were actively seeking treatment for their moderate to severe opioid use disorder.
3. Patients with positive UDS for BPN, barbiturates, or methadone or breath alcohol on the day of check-in to the CRU.
4. Aspartate aminotransferase (AST) levels >3 X the upper limit of normal, alanine aminotransferase (ALT) levels >3 X the upper limit of normal, total bilirubin >1.5 X the upper limit of normal, or creatinine >1.5 X the upper limit of normal on the Screening laboratory assessments and at inpatient check-in, or other clinically significant laboratory abnormalities, which in the opinion of the Investigator may have prevented the patient from safely participating in study.
5. Any clinically significant abnormality on the basis of medical history, vital signs, physical examination, 12-lead electrocardiogram ([ECG], QTcF ≥450 msec for males or ≥470 msec for females), and laboratory evaluation (including hematology, clinical chemistry, urinalysis, and serology [optional]) at Screening, in the opinion of the Investigator.
6. Significant symptoms, medical conditions, or other circumstances which, in the opinion of the Investigator, would have precluded compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may have prevented the patient from safely participating in study (including, but not limited to, the risks described as precautions, warnings, and contraindications in the current version of the Investigator's Brochure for CAM2038).
7. Patients were carefully screened to exclude individuals presenting with a clinically significant history of seizure disorders, history of asthma or other respiratory disorders, head injury, hypertension, or personal history of cardiovascular disease or clinically significant ECG abnormalities.
8. Current diagnosis of Acquired Immune Deficiency Syndrome.
9. Current diagnosis of chronic pain requiring opioids for treatment.
10. Patients who met the criteria for a diagnosis of moderate or severe substance use disorder according to DSM-V criteria for any other substances other than opioids, caffeine, or tobacco.
11. Pregnant or lactating, or planned to become pregnant during the study.
12. Clinically significant history of or current evidence of suicidal ideation or active suicidal behavior as based on the Columbia-Suicide Severity Rating Scale (C-SSRS; grade 4 or 5).
13. Hypersensitivity or allergy to BPN or other opioids or excipients of CAM2038.
14. Intolerance to venipuncture and/or difficulty with venous access, as per the judgment of the Investigator/research staff.
15. Patient was using an investigational drug or monoamine oxidase inhibitor or had used such within the last 30 days (or 5 times the half-life of the drug, if known and longer) prior to first drug administration in the Qualification Phase (i.e., IR morphine sulfate).
16. Required current use of agents that were strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4), such as some azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., clarithromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir).
17. If the patient was currently on probation or had any pending legal action that could have prohibited participation or compliance in the study.
18. A patient who, in the opinion of the Investigator, was considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Walsh, PhD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - New York Psychiatric Institute, New York, New York

REFERENCES:
- [Derived] Bjornsson M, Acharya C, Strandgarden K, Tiberg F. Population Pharmacokinetic Analysis Supports Initiation Treatment and Bridging from Sublingual Buprenorphine to Subcutaneous Administration of a Buprenorphine Depot (CAM2038) in the Treatment of Opioid Use Disorder. Clin Pharmacokinet. 2023 Oct;62(10):1427-1443. doi: 10.1007/s40262-023-01288-6. Epub 2023 Aug 16. PMID 37584841
- [Derived] Walsh SL, Comer SD, Lofwall MR, Vince B, Levy-Cooperman N, Kelsh D, Coe MA, Jones JD, Nuzzo PA, Tiberg F, Sheldon B, Kim S. Effect of Buprenorphine Weekly Depot (CAM2038) and Hydromorphone Blockade in Individuals With Opioid Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):894-902. doi: 10.1001/jamapsychiatry.2017.1874. PMID 28655025

RESULTS

PARTICIPANT FLOW:
Groups:
- CAM2038 q1w, 24 mg: CAM2038 once weekly 24 mg subcutaneous injection will be administered on Day 0 and Day 7. Hydromorphone 0 mg (placebo), 6 mg and 18 mg intramuscular injection will be subsequently administered during 4 challenge sessions on Days 1-3, 4-6, 8-10 and 11-13
- CAM2038 q1w, 32 mg: CAM2038 once weekly 32 mg subcutaneous injection will be administered on Day 0 and Day 7. Hydromorphone 0 mg (placebo), 6 mg and 18 mg intramuscular injection will be subsequently administered during 4 challenge sessions on Days 1-3, 4-6, 8-10 and 11-13
Period: Overall Study
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
Started | 22 | 25
Day 1-3 Hydromorphone Challenge Injs | 22 | 25
Day 4-6 Hydromorphone Challenge Injs | 22 | 24
Day 8-10 Hydromorphone Challenge Injs | 22 | 24
Day11-13 Hydromorphone Challenge Injs | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: A summary of demographics and baseline characteristics will be presented by treatment arm for safety population. The demographic characteristics will consist of age, sex, ethnicity, and race us.
Groups:
- CAM2038 q1w, 24 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo) intramuscular injection will be administered on one day of the 3 days during 4 challenge sessions on Days 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 32 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo) intramuscular injection will be administered on one day of the 3 days during 4 challenge sessions on Days 1-3, 4-6, 8-10 and 11-13.
- Total: Total of all reporting groups
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.3) | 35.6 (9.1) | 35.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 15 | 24
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
BMI, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (4.28) | 24.4 (4.25) | 24.8 (4.24)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase Drug Liking Visual Analog Scale (VAS) Emax Scores for Baseline and Four Challenge Sessions Compared to Baseline (Completer Population) for CAM2038 q1w, 24 mg
Description: Treatment Phase Drug Liking Visual Analog Scale (VAS) item "At this moment, my liking of this drug is" for Baseline and Four Challenge sessions Compared to Baseline (Completer Population) for CAM2038 q1w, 24 mg, where values can range from 0 (strong disliking) to 100 (strong liking) and 50 is the neutral point. Higher scores mean worse outcome.
Time Frame: 17 days
Population: Mean Drug Liking VAS Scores over Time for CAM2038 q1w 24 mg by Hydromorphone Challenge Session, Completer Population (N=22)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- CAM2038 q1w, 24 mg - Hydromorphone 0 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo) intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 24 mg - Hydromorphone 6 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 6 mg intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 24 mg - Hydromorphone 18 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 18 mg intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
Arm/Group | CAM2038 q1w, 24 mg - Hydromorphone 0 mg | CAM2038 q1w, 24 mg - Hydromorphone 6 mg | CAM2038 q1w, 24 mg - Hydromorphone 18 mg
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  Baseline | 50.6 (1.48) | 83.2 (1.48) | 92.7 (1.48)
  Days 1-3 | 51.3 (0.84) | 52.2 (0.84) | 53.1 (0.84)
  Days 4-6 | 50.8 (0.84) | 52.1 (0.84) | 58.3 (0.84)
  Days 8 -10 | 51.1 (0.84) | 52.6 (0.84) | 52.9 (0.84)
  Days 11-13 | 51.0 (0.84) | 51.9 (0.84) | 54.6 (0.84)

2. Primary Outcome: Treatment Phase Drug Liking Visual Analog Scale (VAS) Maximum Effect (Emax) Scores for Baseline and Four Challenge Sessions Compared to Baseline (Completer Population) for CAM2038 q1w, 32 mg
Description: Treatment Phase Drug Liking Visual Analog Scale (VAS) item "At this moment, my liking of this drug is" for Baseline and Four Challenge sessions Compared to Baseline (Completer Population), where values can range from 0 (strong disliking) to 100 (strong liking) and 50 is the neutral point. Higher scores mean worse outcome.
Time Frame: 17 days
Population: Mean Drug Liking VAS Scores over Time for CAM2038 q1w 32 mg by Hydromorphone Challenge Session, Completer Population (N=24)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- CAM2038 q1w, 32 mg - Hydromorphone 0 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo) intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 32 mg - Hydromorphone 6 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 6 mg intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 32 mg - Hydromorphone 18 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 18 mg intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
Arm/Group | CAM2038 q1w, 32 mg - Hydromorphone 0 mg | CAM2038 q1w, 32 mg - Hydromorphone 6 mg | CAM2038 q1w, 32 mg - Hydromorphone 18 mg
Number analyzed (Participants) | 24 | 24 | 24
units on a scale
  Baseline | 52.9 (1.70) | 79.6 (1.70) | 93.2 (1.70)
  Days 1-3 | 51.6 (1.01) | 52.5 (1.01) | 54.0 (1.01)
  Days 4-6 | 51.5 (1.01) | 53.0 (1.01) | 56.0 (1.01)
  Days 8 -10 | 51.7 (1.01) | 52.3 (1.01) | 54.2 (1.01)
  Days 11-13 | 51.2 (1.01) | 52.1 (1.01) | 54.8 (1.01)

3. Primary Outcome: Inferential Analysis Results Drug Liking Visual Analog Scale (VAS) for Maximum Effect (Emax) Scores for Qualification/Baseline and Four Challenge Sessions (Completer Population) for CAM2038 q1w, 24 mg
Description: Inferential Analysis Results Drug Liking Visual Analog Scale (VAS) item "At this moment, my liking of this drug is" for Qualification/Baseline and Four Challenge sessions (Completer Population) for CAM2038 q1w, 24 mg, where values can range from 0 (strong disliking) to 100 (strong liking) and 50 is the neutral point. Higher scores mean worse outcome.
Time Frame: 17 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- CAM2038 q1w, 24 mg - Hydromorphone 6 Mg-Hydromorphone 0 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo) and 6 mg intramuscular injection will be administered on 2 of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 24 mg - Hydromorphone 18 mg- Hydromorphone 0mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 18 mg and Hydromorphone 0 mg intramuscular injection will be administered on 2 of the 3 days during baseline and 4 challenge sessions on Days -3--1,1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 24 mg - Hydromorphone 18 mg- Hydromorphone 6 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 18 mg and Hydromorphone 6 mg intramuscular injection will be administered on 2 of the 3 days during baseline and 4 challenge sessions on Days -3--1,1-3, 4-6, 8-10 and 11-13.
Arm/Group | CAM2038 q1w, 24 mg - Hydromorphone 6 Mg-Hydromorphone 0 mg | CAM2038 q1w, 24 mg - Hydromorphone 18 mg- Hydromorphone 0mg | CAM2038 q1w, 24 mg - Hydromorphone 18 mg- Hydromorphone 6 mg
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  Qualification/Baseline | 32.7 (1.90) | 42.1 (1.90) | 9.5 (1.90)
  Days 1-3 | 0.9 (1.12) | 1.8 (1.12) | 0.9 (1.12)
  Days 4-6 | 1.3 (1.12) | 7.4 (1.12) | 6.2 (1.12)
  Days 8 -10 | 1.5 (1.12) | 1.8 (1.12) | 0.3 (1.12)
  Days 11-13 | 0.9 (1.12) | 3.6 (1.12) | 2.7 (1.12)

4. Primary Outcome: Inferential Analysis Results Drug Liking Visual Analog Scale (VAS) Maximum Effect (Emax) Scores for Qualification/Baseline and Four Challenge Sessions (Completer Population) for CAM2038 q1w, 32 mg
Description: Inferential Analysis Results Drug Liking Visual Analog Scale (VAS) item "At this moment, my liking of this drug is" for Qualification/Baseline and Four Challenge sessions (Completer Population) for CAM2038 q1w, 32 mg, where values can range from 0 (strong disliking) to 100 (strong liking) and 50 is the neutral point. Higher scores mean worse outcome.
Time Frame: 17 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- CAM2038 q1w, 32 mg - Hydromorphone 6 Mg-Hydromorphone 0 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo) and 6 mg intramuscular injection will be administered on 2 of the 3 days during baseline and 4 challenge sessions on Days -3--1,1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 32 mg - Hydromorphone 18 mg- Hydromorphone 0mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 18 mg and Hydromorphone 0 mg intramuscular injection will be administered on 2 of the 3 days during baseline and4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 32 mg - Hydromorphone 18 mg- Hydromorphone 6 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 18 mg and Hydromorphone 6 mg intramuscular injection will be administered on 2 of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
Arm/Group | CAM2038 q1w, 32 mg - Hydromorphone 6 Mg-Hydromorphone 0 mg | CAM2038 q1w, 32 mg - Hydromorphone 18 mg- Hydromorphone 0mg | CAM2038 q1w, 32 mg - Hydromorphone 18 mg- Hydromorphone 6 mg
Number analyzed (Participants) | 24 | 24 | 24
units on a scale
  Qualification/Baseline | 26.7 (2.40) | 40.3 (2.40) | 13.7 (2.40)
  Days 1-3 | 0.9 (1.05) | 2.4 (1.05) | 1.5 (1.05)
  Days 4-6 | 1.5 (1.05) | 4.5 (1.05) | 3.0 (1.05)
  Days 8 -10 | 0.5 (1.05) | 2.5 (1.05) | 2.0 (1.05)
  Days 11-13 | 1.0 (1.05) | 3.6 (1.05) | 2.6 (1.05)

5. Secondary Outcome: Inferential Analysis Results for Unipolar High Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population)
Description: Inferential Analysis Results for Unipolar High Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population) comparing hydromorphone challenge doses in each of the baseline and four challenge sequence with each other, presented as Least Squares (LS) Mean with Standard Error (SE) and 95% Confidence Interval (CI). VAS item "At this moment, I feel high" where values can range from 0 (Not at all High) to 100 (Extremely High).
Time Frame: 15 days
Population: Completer Population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- CAM2038 q1w, 24 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7.
- CAM2038 q1w, 32 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7.
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
Number analyzed (Participants) | 22 | 24
units on a scale
  Baseline HMO 6mg-HMO 0mg | 62.4 [53.7 to 71.2] | 47.3 [35.8 to 58.7]
  Baseline HMO18mg-HMO 0 mg | 84.6 [75.8 to 93.3] | 77.0 [65.5 to 88.4]
  Baseline HMO 18mg - HMO 6mg | 22.2 [13.4 to 30.9] | 29.7 [18.3 to 41.2]
  Challenge Session 1 HMO 6mg - HMO 0mg | 4.3 [-0.4 to 9.0] | 3.1 [-0.4 to 6.6]
  Challenge Session 1 HMO 18mg - HMO 0mg | 3.6 [-1.1 to 8.3] | 3.2 [-0.3 to 6.7]
  Challenge Session 1 HMO 18mg-HMO 6mg | -0.8 [-5.4 to 3.9] | 0.1 [-3.4 to 3.6]
  Challenge Session 2 HMO 6mg - HMO 0mg | 1.8 [-2.9 to 6.5] | 1.5 [-2.0 to 5.1]
  Challenge Session 2 HMO 18mg - HMO 0mg | 15.3 [10.6 to 20.0] | 6.5 [3.0 to 10.1]
  Challenge Session 2 HMO 18mg - HMO 6mg | 13.5 [8.8 to 18.2] | 5.0 [1.5 to 8.6]
  Challenge Session 3 HMO6mg - HMO 0mg | 2.6 [-2.1 to 7.2] | 0.9 [-2.6 to 4.5]
  Challenge Session 3 HMO 18mg - HMO 0mg | 3.9 [-0.8 to 8.5] | 5.4 [1.9 to 9.0]
  Challenge Session 3 HMO 18mg - HMO 6mg | 1.3 [-3.4 to 6.0] | 4.5 [1.0 to 8.1]
  Challenge Session 4 HMO 6mg - HMO 0mg | 2.1 [-2.6 to 6.8] | 1.3 [-2.2 to 4.8]
  Challenge Session 4 HMO 18mg - HMO 0mg | 6.4 [1.7 to 11.0] | 6.0 [2.4 to 9.5]
  Challenge Session 4 HMO 18mg - HMO 6mg | 4.2 [-0.4 to 8.9] | 4.7 [1.1 to 8.2]

6. Secondary Outcome: Inferential Analysis Results for Unipolar Good Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population)
Description: Inferential Analysis Results for Unipolar Good Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population) comparing hydromorphone challenge doses in each of the baseling and four challenge sequences with each other, presented as Least Squares (LS) Mean with Standard Error (SE) and 95% Confidence Interval (CI). VAS item "At this moment, I feel good drug effects" where values can range from 0 (Not at all ) to 100 (Extremely).
Time Frame: 15 days
Population: Completer Population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
Number analyzed (Participants) | 22 | 24
units on a scale
  Baseline HMO 6mg-HMO 0mg | 61.6 [52.5 to 70.7] | 52.8 [43.3 to 62.3]
  Baseline HMO 18mg-HMO 0mg | 85.4 [76.4 to 94.5] | 81.8 [72.3 to 91.4]
  Baseline HMO18mg-HMO 6mg | 23.9 [14.8 to 32.9] | 29.1 [19.6 to 38.6]
  Challenge Session 1 HMO 6mg - HMO 0mg | 0.8 [-5.1 to 6.6] | 2.8 [-1.1 to 6.7]
  Challenge Session 1 HMO 18mg - HMO 0mg | 1.3 [-4.5 to 7.2] | 4.9 [1.0 to 8.8]
  Challenge Session 1 HMO 18mg-HMO 6mg | 0.6 [-5.3 to 6.4] | 2.1 [-1.8 to 6.0]
  Challenge Session 2 HMO 6mg - HMO 0mg | 1.8 [-4.0 to 7.7] | 1.7 [-2.2 to 5.6]
  Challenge Session 2 HMO 18mg - HMO 0mg | 15.8 [10.0 to 21.7] | 7.3 [3.4 to 11.2]
  Challenge Session 2 HMO18mg - HMO 6mg | 14.0 [8.1 to 19.8] | 5.6 [1.7 to 9.5]
  Challenge Session 3 HMO6mg - HMO 0mg | 2.4 [-3.4 to 8.2] | 0.8 [-3.1 to 4.7]
  Challenge Session 3 HMO 18mg - HMO 0mg | 4.7 [-1.2 to 10.5] | 4.9 [1.0 to 8.9]
  Challenge Session 3 HMO 18mg - HMO 6mg | 2.3 [-3.5 to 8.1] | 4.1 [0.2 to 8.1]
  Challenge Session 3 HMO 6mg - HMO 0mg | 2.2 [-3.6 to 8.0] | 0.7 [-3.2 to 4.7]
  Challenge Session 4 HMO 18mg - HMO 0mg | 7.1 [1.3 to 13.0] | 6.0 [2.1 to 9.9]
  Challenge Session 4 HMO 18mg - HMO 6mg | 4.9 [-0.9 to 10.8] | 5.2 [1.3 to 9.2]

7. Secondary Outcome: Analysis of Treatment Phase Unipolar Bad Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) in 24 mg CAM2038 q1w Group (Completer Population)
Description: Analysis of Treatment Phase Unipolar Bad Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) in 24 mg CAM2038 q1w group (Completer Population) , presented as Least Squares (LS) mean with Standard Error (SE) for all 3 doses of hydromorphone in baseline and 4 Challenge Sessions. VAS item "At this moment, I feel bad effects" where values can range from 0 (Not at all) to 100 (Extremely).
Time Frame: 15 days
Population: Completer Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- CAM2038 q1w, 24 mg - Hydromorphone 0 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0mg (placebo) intramuscular injection will be administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
Arm/Group | CAM2038 q1w, 24 mg - Hydromorphone 0 mg | CAM2038 q1w, 24 mg - Hydromorphone 6 mg | CAM2038 q1w, 24 mg - Hydromorphone 18 mg
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  Baseline | 3.0 (3.18) | 8.4 (3.18) | 13.1 (3.18)
  Challenge Session 1 (Days 1-3) | 5.0 (1.17) | 0.9 (1.17) | 0.8 (1.17)
  Challenge Session 2 (Days 4-6) | 1.5 (1.17) | 0.8 (1.17) | 1.6 (1.17)
  Challenge Session 3 (Days 8-10) | 0.8 (1.17) | 0.7 (1.17) | 1.6 (1.17)
  Challenge Session 4 (Days 11-13) | 1.0 (1.17) | 1.0 (1.17) | 0.9 (1.17)

8. Secondary Outcome: Analysis of Treatment Phase Unipolar Bad Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) in 32 mg CAM2038 q1w Group (Completer Population)
Description: Analysis of Treatment Phase Unipolar Bad Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) in 32 mg CAM2038 q1w group (Completer Population) , presented as Least Squares (LS) mean with Standard Error (SE) for all 3 doses of hydromorphone in baseline and 4 Challenge Sessions. VAS item "At this moment, I feel bad effects" where values can range from 0 (Not at all) to 100 (Extremely).
Time Frame: 15 days
Population: Completer Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CAM2038 q1w, 32 mg - Hydromorphone 0 mg | CAM2038 q1w, 32 mg - Hydromorphone 6 mg | CAM2038 q1w, 32 mg - Hydromorphone 18 mg
Number analyzed (Participants) | 24 | 24 | 24
units on a scale
  Baseline | 5.9 (3.47) | 13.1 (3.47) | 12.6 (3.47)
  Challenge Session 1 (Days 1-3) | 1.2 (0.67) | 1.3 (0.67) | 1.4 (0.67)
  Challenge Session 2 (Days 4-6) | 0.5 (0.67) | 1.4 (0.67) | 2.1 (0.67)
  Challenge Session 3 (Days 8-10) | 0.6 (0.67) | 0.8 (0.67) | 2.8 (0.67)
  Challenge Session 4 (Days 11-13) | 0.6 (0.67) | 1.0 (0.67) | 1.3 (0.67)

9. Secondary Outcome: Analysis Results for Unipolar Desire to Use Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population)
Description: Analysis Results for Desire to Use Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population) comparing hydromorphone challenge doses in each of the baseline and four challenge sequence with each other, presented as Least Squares (LS) Mean with Standard Error (SE) and 95% Confidence Interval (CI). VAS item "At this moment, I desire opiods" where values can range from 0 (Definitely not) to 100 (Definitely so).
Time Frame: 15 days
Population: (Completer Population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
Number analyzed (Participants) | 22 | 24
units on a scale
  Baseline HMO 6mg-HMO 0mg | -18.0 (4.50) | 14.1 (3.76)
  Baseline HMO 18mg-HMO 0mg | -31.0 (4.50) | -29.2 (3.75)
  Baseline HMO18mg-HMO 6mg | 013.0 (4.50) | -15.1 (3.75)
  Challenge Session 1 HMO 6mg - HMO 0mg | -0.2 (4.03) | 8.7 (5.09)
  Challenge Session 1 HMO 18mg - HMO 0mg | 1.8 (4.03) | -5.7 (5.08)
  Challenge Session 1 HMO 18mg-HMO 6mg | 2.0 (4.03) | -14.4 (5.08)
  Challenge Session 2 HMO 6mg - HMO 0mg | -3.8 (4.03) | -3.1 (5.09)
  Challenge Session 2 HMO 18mg - HMO 0mg | -6.2 (4.03) | 0.7 (5.08)
  Challenge Session 2 HMO 18mg - HMO 6mg | -2.4 (4.03) | 3.7 (5.08)
  Challenge Session 3 HMO6mg - HMO 0mg | -2.8 (4.03) | 2.2 (5.09)
  Challenge Session 3 HMO 18mg - HMO 0mg | -1.8 (4.03) | 0.4 (5.08)
  Challenge Session 3 HMO 18mg - HMO 6mg | 1.0 (4.03) | -1.8 (5.08)
  Challenge Session 4 HMO 6mg - HMO 0mg | -2.2 (4.03) | -0.2 (5.09)
  Challenge Session 4 HMO 18mg - HMO 0mg | -4.5 (4.03) | 0.9 (5.08)
  Challenge Session 4 HMO 18mg - HMO 6mg | -2.3 (4.03) | 1.1 (5.08)

10. Secondary Outcome: Analysis Results for Bipolar Alertness/Drowsiness Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population)
Description: Analysis Results for Bipolar Alertness/Drowsiness Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population) presented as Least Squares (LS) mean with Standard Error (SE) for all 3 doses of hydromorphone in baseline and 4 Challenge Sessions. VAS item "At this moment, my mental state is" where values can range from 0 (Very Drowsy) to 100 (Very alert), with 50 being neutral (Neither drowsy nor alert).
Time Frame: 15 days
Population: (Completer Population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
Number analyzed (Participants) | 22 | 24
units on a scale
  Baseline HMO 6mg-HMO 0mg | -18.0 (4.5) | -14.1 (3.76)
  Baseline HMO 18mg-HMO 0mg | -31.0 (4.50) | -29.2 (3.75)
  Baseline HMO18mg-HMO 6mg | -13.0 (4.50) | -15.1 (3.75)
  Challenge Session 1 HMO 6mg - HMO 0mg | -2.2 (3.89) | 1.7 (3.05)
  Challenge Session 1 HMO 18mg - HMO 0mg | -4.9 (3.89) | -0.8 (3.05)
  Challenge Session 1 HMO 18mg-HMO 6mg | -2.8 (3.89) | -2.5 (3.05)
  Challenge Session 2 HMO 6mg - HMO 0mg | -6.2 (3.89) | -2.0 (3.05)
  Challenge Session 2 HMO 18mg - HMO 0mg | -8.3 (3.89) | -2.7 (3.05)
  Challenge Session 2 HMO 18mg - HMO 6mg | -2.1 (3.89) | -0.7 (3.05)
  Challenge Session 3 HMO6mg - HMO 0mg | -0.2 (3.89) | -0.9 (3.05)
  Challenge Session 3 HMO 18mg - HMO 0mg | -7.5 (3.89) | -4.3 (3.05)
  Challenge Session 3 HMO 18mg - HMO 6mg | -7.4 (3.89) | -3.4 (3.05)
  Challenge Session 4 HMO 6mg - HMO 0mg | 0.7 (3.89) | 1.8 (3.05)
  Challenge Session 4 HMO 18mg - HMO 0mg | -2.1 (3.89) | -0.2 (3.05)
  Challenge Session 4 HMO 18mg - HMO 6mg | -2.8 (3.89) | -2.0 (3.05)

11. Secondary Outcome: Analysis Results for Unipolar Any Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population)
Description: Analysis Results for Unipolar Any Drug Effects Visual Analog Scale (VAS) for Maximum Effect (Emax) (Completer Population) presented as Least Squares (LS) mean with Standard Error (SE) for all 3 doses of hydromorphone in baseline and 4 Challenge Sessions. VAS item "At this moment, I fell any drug effects" where values can range from 0 (Not at all) to 100 (Extremely).
Time Frame: 15 days
Population: (Completer Population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
Number analyzed (Participants) | 22 | 24
units on a scale
  Baseline HMO 6mg-HMO 0mg | 63.2 (4.49) | 47.8 (5.25)
  Baseline HMO 18mg-HMO 0mg | 83.9 (4.49) | 76.4 (5.24)
  Baseline HMO18mg-HMO 6mg | 20.7 (4.49) | 28.6 (5.24)
  Challenge Session 1 HMO 6mg - HMO 0mg | 4.0 (2.27) | 3.2 (2.36)
  Challenge Session 1 HMO 18mg - HMO 0mg | 3.5 (2.27) | 6.8 (2.35)
  Challenge Session 1 HMO 18mg-HMO 6mg | -0.5 (2.27) | 3.6 (2.35)
  Challenge Session 2 HMO 6mg - HMO 0mg | 1.6 (2.27) | 3.6 (2.36)
  Challenge Session 2 HMO 18mg - HMO 0mg | 13.6 (2.27) | 5.9 (2.35)
  Challenge Session 2 HMO 18mg - HMO 6mg | 11.9 (2.27) | 2.2 (2.35)
  Challenge Session 3 HMO6mg - HMO 0mg | 2.4 (2.27) | -1.1 (2.36)
  Challenge Session 3 HMO 18mg - HMO 0mg | 4.6 (2.27) | 3.3 (2.35)
  Challenge Session 3 HMO 18mg - HMO 6mg | 2.2 (2.27) | 4.4 (2.35)
  Challenge Session 4 HMO 6mg - HMO 0mg | 1.5 (2.27) | -1.1 (2.36)
  Challenge Session 4 HMO 18mg - HMO 0mg | 6.9 (2.27) | 2.1 (2.35)
  Challenge Session 4 HMO 18mg - HMO 6mg | 5.4 (2.27) | 3.2 (2.35)

ADVERSE EVENTS:
Time Frame: All AEs were documented and followed from the time the patient had signed the informed consent form until 14 days after the Follow-up Visit (or 30 days after Early Termination). The maximum number of days being 61 days.
Groups:
- CAM2038 q1w, 24 mg: CAM2038 q1w 24 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo), 6 mg, and 18 mg intramuscular injections each being administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
- CAM2038 q1w, 32 mg: CAM2038 q1w 32 mg will be administered by subcutaneous injection on Day 0 and Day 7. Hydromorphone 0 mg (placebo), 6 mg, and 18 mg intramuscular injections each being administered on one day of the 3 days during baseline and 4 challenge sessions on Days -3--1, 1-3, 4-6, 8-10 and 11-13.
Arm/Group | CAM2038 q1w, 24 mg | CAM2038 q1w, 32 mg
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 13/22 | 24/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAM2038 q1w, 24 mg (N=22) | CAM2038 q1w, 32 mg (N=25)
Constipation (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 1 | 3
Faeces Hard (Gastrointestinal disorders) | 0 | 2
Injection Site Pain (General disorders) | 2 | 3
Injection Site Erythema (General disorders) | 2 | 2
Injection Site Pruritus (General disorders) | 1 | 2
Injection site Haemorrhage (General disorders) | 0 | 2
Dermatitis Contac (Skin and subcutaneous tissue disorders) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT02611752/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02611752/SAP_001.pdf